CLINICAL TRIAL: NCT05080205
Title: Effects of Morbid Obesity and Bariatric Surgery on Brain Inflammation, Insulin Resistance and Activation of Central Reward System Studied Using PET- and MRI-imaging
Brief Title: Effects of Morbid Obesity and Bariatric Surgery on Brain Inflammation, Insulin Resistance and Central Reward System
Acronym: BariBrainPET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Pirjo Nuutila, professor, Turku University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BariBrain-PET; T153/2018 (Other: The Hospital District of Southwest Finland)
Record Dates: First submitted 2018-06-06; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Obesity, Morbid; Insulin Resistance
Keywords: obesity; insulin resistance; central nervous system inflammation; bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Insulin Resistance; Obesity | interventions — Bariatric Surgery; Gastric Bypass

STUDY DESIGN:
Intervention Model Description: 60 subjects undergoing bariatric surgery (either Roux-en-Y gastric bypass or Sleeve gastrectomy) and 30 healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morbidly obese subjects (Experimental): Bariatric surgery (Roux-en-Y gastric bypass or sleeve gastrectomy)
  Interventions: Procedure: Bariatric surgery
- Control subjects (No Intervention): Non-obese controls are only studied at baseline

INTERVENTIONS:
Procedure: Bariatric surgery — Roux-en-Y gastric bypass or sleeve gastrectomy, chosen based on routine evaluation process
  Other Names: Roux-en-Y gastric bypass; Sleeve gastrectomy
  Arms: Morbidly obese subjects

SUMMARY:
Background: Morbid obesity is associated with decreased brain µ-opioid receptor availability, possibly resulting in higher food intake needed to gain pleasure from eating. This decrease seems to normalize already 6 months after bariatric surgery, but the longer-term effects have not been studied. Obesity and insulin resistance result in significantly increased brain insulin-stimulated glucose uptake, whereas in every other tissue glucose uptake is lower. One possible explanation to this could be central inflammation and activation of brain glial cells, which has been shown to occur in animal models of obesity. Obesity has also been shown to associate with increased risk of Alzheimer's disease and cognitive decline in several studies.

Aims: The first objective of this study is to both study the effects of bariatric surgery as well as compare the effects of gastric bypass and sleeve gastrectomy on food-associated pleasure, extending the follow-up period to 2 years postoperatively. The second aim is to investigate the effect of morbid obesity and weight loss on brain inflammation and gliosis and its association with increased brain insulin-stimulated glucose uptake. Furthermore, association of obesity, insulin resistance, central inflammation and neurocognitive dysfunction are evaluated.

DETAILED DESCRIPTION:
Methods: A total of 60 morbidly obese subjects, 30 assigned for Roux-en-Y gastric bypass and 30 for sleeve gastrectomy according to routine treatment protocols will be recruited for this study. A control group of 30 healthy subjects will also be recruited. We will perform 1) structural MRI and MRS, 2) functional MRI during tasting and visual food cues, 3) PET imaging of µ-opioid receptor availability using [11C]-carfentanil, 4) PET imaging of cerebral inflammation and astrocyte activation using [11C]-PK11195, 5) measurement of whole-body and tissue insulin sensitivity by combining hyperinsulinemic, euglycemic clamp with [18F]-FDG-PET, 6) neuropsychological testing. The control group will only be studied once, whereas study procedures will be repeated for the morbidly obese before very-low calorie diet and 6, 12 and 24 months postoperatively.

ELIGIBILITY:
Inclusion criteria:

Morbidly obese group

1. BMI 35.0-45.0 kg/m2, or BMI 32.0-45.0 kg/m2 and diagnosed diabetes
2. Age 18-60 years
3. Eligible to bariatric surgery evaluated according to normal treatment paradigm

Non-obese controls

1. BMI 18-27 kg/m2
2. Age 18-60 years
3. Fasting plasma glucose ≤6.1 mmol/L
4. Normal values in 2-hour oral glucose tolerance test

Exclusion criteria:

Morbidly obese group

1. Metal objects in the body (including pacemakers, metallic artificial valve prostheses, inner ear implants, surgical clipses, braces, foreign fragments)
2. Previous participation in PET studies
3. Pregnancy
4. Poor compliance, alcohol or drug abuse
5. Weight over 150 kg or waist circumference over 150 cm
6. Diabetes with fasting glucose levels ≥7.0 mmol/L, or treatment with insulin
7. Any chronic disease, medication or condition that could create a hazard to subject safety, endanger study procedures or interfere with the interpretation of results.

Non-obese controls

1. Metal objects in the body (including pacemakers, metallic artificial valve prostheses, inner ear implants, surgical clipses, braces, foreign fragments)
2. Previous participation in PET studies
3. Pregnancy
4. Poor compliance, alcohol or drug abuse
5. Smoking
6. History of eating disorders, drastic weight-gain or weight-loss
7. History of psychiatric disorders
8. Any chronic disease, medication or condition that could create a hazard to subject safety, endanger study procedures or interfere with the interpretation of results

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in central inflammation | Controls: 0 months; Morbidly obese: preoperatively, 6 months postoperatively
  Assessment of brain glial cell activation using [11C]-PK11195 tracer and positron emission tomography

SECONDARY OUTCOMES:
Changes in central reward system using fMRI imaging | Controls: 0 months; Morbidly obese: preoperatively, 6 months, 12 months, 24 months postoperatively
  Assessment of brain reward system activation after visual/taste cues using functional MRI
Changes in brain μ-opioid receptor availability using PET imaging | Controls: 0 months; Morbidly obese: preoperatively, 6 months, 12 months postoperatively
  Assessment of brain μ-opioid receptor availability using [11C]-carfentanil tracer and positron emission tomography
Changes in cognitive function studied with testing | Controls: 0 months; Morbidly obese: preoperatively, 6 months, 12 months, 24 months postoperatively
  Neuropsychological testing focusing on memory, decision-making and inhibition
Changes in whole-body insulin sensitivity usign FDG-PET imaging | Controls: 0 months; Morbidly obese: preoperatively, 6 months postoperatively
  Assessment of whole-body insulin sensitivity using hyperinsulinemic, euglycemic clamp
Changes in tissue-specific insulin sensitivity using FDG-PET imaging | Controls: 0 months; Morbidly obese: preoperatively
  Assessment of insulin-stimulated glucose uptake in the brain, liver, skeletal muscle and adipose tissue by performing positron emission tomography with [18F]-fluorodeoxyglucose tracer during hyperinsulinemic, euglycemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Nuutila, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: Yes
Under preparation.
Supporting Information: Study Protocol, SAP, ICF, CSR